## Official title of the study:

Pathophysiological Mechanisms Elicited by Ischemia and Metabolic Co-morbidities in Myocardium of Patients with Coronary Artery Disease

**NCT** number:

NCT03179137

**Document date:** 

June 16, 2020

## **Participating institutions:**

University of Split School of Medicine
University Hospital of Split





## STUDY PROTOCOL

**Study location:** Clinic for Cardiovascular diseases and Department of Cardiac Surgery, University Hospital of Split

**Ethical Approval:** This study protocol had been reviewed and approved by the Ethics Committees of the University of Split School of Medicine and University Hospital of Split.

**Patient recruitment:** All patients fulfilling the inclusion criteria will receive a printed material containing information regarding the study and any potential questions will be answered by the recruiting personnel. A signed informed consent form will be a prerequisite for patient inclusion into the study.

## **Study protocol:**

